CLINICAL TRIAL: NCT05633576
Title: Steroid Eye Drops Versus Placebo Eye Drops in Chronic Central Serous Chorioretinopathy Trial (PICS Trial)
Brief Title: Steroid Eye Drops in Chronic Central Serous Chorioretinopathy
Acronym: PICS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Oogziekenhuis Rotterdam (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 112907
Record Dates: First submitted 2022-11-21; First posted 2022-12-01 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Chronic Central Serous Chorioretinopathy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- steroid eye drops (Active Comparator): In this treatment arm, patients will self-administer the steroid eye drops three times a day for four consecutive weeks.
  Interventions: Drug: steroid eye drops
- Placebo (Placebo Comparator): In this treatment arm, patients will self-administer the placebo eye drops three times a day for four consecutive weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: steroid eye drops — Self-administration of steroid eye drops three times a day for four consecutive weeks.
  Arms: steroid eye drops
Drug: Placebo — Self-administration of placebo eye drops three times a day for four consecutive weeks.
  Arms: Placebo

SUMMARY:
In this pilot study the effect and safety of the use of steroid eye drops in chronic central serous chorioretinopathy (cCSC) will be evaluated. The study is conducted as a randomized single-blind placebo-controlled trial. Forty patients will be randomized to either steroid eye drops or placebo eye drops. Patients will self-administer the eye drops three times a day for four weeks.

DETAILED DESCRIPTION:
Severe chronic central serous chorioretinopathy (cCSC) is a disease part of the pachychoroid disease spectrum and is characterized by the presence of subretinal and intraretinal fluid. Left untreated these patients are at serious risk of irreversible vision loss. The most effective treatment is photodynamic therapy (PDT), which is expensive, invasive and currently only available to a limited extent. Pachychoroid diseases are correlated to the use of systemic steroids or an increase in cortisol, to stress, sleep apnea and sildenafil use. In many cases there is no clear correlation to one of the risk factors. However, in clinical practice, a strikingly good effect on sub- and intraretinal fluid in another disease that is part of the pachychoroid disease spectrum was seen by using steroid eye drops (PPS; peripapillary pachychoroid disease). Steroid eye drops are used in many ophthalmic diseases, however, there is no clinical experience for the use steroid eye drops in cCSC.

The aim of this study is to assess the safety and the effect of steroid eye drops in patients suffering from cCSC for clinical, multimodal imaging, anatomical and functional outcomes. In addition, we want to gain insight in the mechanism of action and to investigate the effect of topical steroids on the intraocular pressure.

No previous studies have evaluated the effect of steroid eye drops on cCSC, therefore this study is set up as a pilot study, with a randomized, single-blinded, placebo controlled trial design. In total, forty patients will be randomized to either steroid eye drops or placebo eye drops. Patients will self-administer the eye drops three times a day for four weeks. The study will last for four weeks per patient and each patient will visit the outpatient clinic 2 times.

Treatment response will be objectified by multimodal imaging and by measuring the best-corrected visual acuity, after four weeks of using steroid eye drops or placebo.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: All patients will undergo multimodal imaging before inclusion and at the end point of the study, this includes invasive studies. All studies are part of the regular clinical work-up for cCSC and no additional (invasive) investigations will be performed. The use of steroid eye drops holds the risk of an increasement of intraocular pressure (IOP) and may induce cataract. However, both these risks are neglectable when used for 4 weeks only and outweighs the possible reductive effect of steroid eye drops on subretinal and intraretinal fluid.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 18 years or older
* Subretinal and/or intraretinal fluid on OCT and subjective visual loss or presence of Subretinal and/or intraretinal fluid for 3 months or longer
* Patient is able to self-administer eye drops
* Complex or Severe Chronic Central Serous Chorioretinopathy, with at least one of the following clinical findings that are present within the vascular arcades: Cumulative areas (>2 optic disc diameters) of diffuse atrophic RPE alterations visualized on mid-phase FA or on FAF; Multifocal "hot spots": at least 2 "hot spots" of leakage separated by at least 1 disc diameter of nonhyperfluorescent healthy-appearing retina on mid-phase FA; Diffuse leakage: an area of diffuse fluorescein leakage >1 optic disc diameter on mid-phase FA, without an evident leaking focus; Presence of posterior cystoid retinal degeneration assessed on OCT.

Exclusion Criteria:

* Evidence of other retinal diagnoses: ((History of) exudative age-related macular degeneration, Suspicion of secondary choroidal neovascularization, Polypoidal choroidal vasculopathy, Multifocal choroiditis, Retinal vascular occlusions, Pseudoxanthoma elasticum, Amblyopia, Severe myopia (more than -6 diopters).
* Current treatment with corticosteroids or corticosteroid use within 3 months before the baseline visit
* Treatment with PDT, subthreshold micropulse laser or focal laser photocoagulation 6 months prior to the baseline visit.
* Treatment with anti-vascular endothelial growth factor (anti-VEGF), MR-antagonists or carbonic anhydrase inhibitors within 6 weeks prior to the baseline visit. If patients were treated with anti-VEGF, MR-antagonists or carbonic anhydrase inhibitors 3 months to 6 weeks prior to the baseline, patients will only be included if there was no sufficient response to treatment.
* Pregnant or breastfeeding women
* Allergy to topical ophthalmic steroids.
* Media opacities that prohibit detailed multimodal imaging
* (BCVA <20/200) (Snellen equivalent)
* Contraindications for fluorescein angiography or ICG angiography (known allergies especially against shellfish, previous reactions)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-02-19 (Actual); Primary Completion 2025-06-19 (Estimated); Study Completion 2025-07-19 (Estimated)

PRIMARY OUTCOMES:
Change in sub- and intraretinal fluid on OCT scan | 1 month after the start of treatment
  The primary outcome measure of this study is the effect of steroid eye drops in cCSC on the amount of sub and intraretinal fluid. The difference in the amount of sub- and intraretinal fluid will be compared between the OCT scan made prior to the study and the OCT scan made at the second consultation after the study medication has been used for four weeks.

SECONDARY OUTCOMES:
Change in best corrected visual acuity | 1 month after the start of treatment
  Mean change in BCVA between baseline and after using the study medication for 4 weeks.
Intra ocular pressure (IOP) | 1 month after the start of treatment
  Mean change in IOP between baseline and after using the study medication for 4 weeks.
Change of hyperfluorescent areas on fluorescence angiography (FA) | 1 month after the start of treatment
  Mean change in hyperfluorescent areas on FA between baseline and after using the study medication for 4 weeks.
Change of hypercyanescent areas on Indocyanine Green Angiography (ICGA) | 1 month after the start of treatment
  Mean change in hypercyanescent areas on ICGA between baseline and after using the study medication for 4 weeks.

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Radboud University Medical Center, Nijmegen
  - Rotterdam Eye Hospital, Rotterdam

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD